CLINICAL TRIAL: NCT05945615
Title: Evaluation of Ophthalmic Oxymetazoline as an Adjunct Treatment for Acquired Blepharoptosis Due to Periocular Synkinesis.
Brief Title: Oxymetazoline Drops for Acquired Blepharoptosis From Synkinesis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jessyka Lighthall, Chief, Facial Plastic and Reconstructive Surgery, Associate Professor, Department of Otolaryngology-Head and Neck Surgery, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00022691
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-04

CONDITIONS: Blepharoptosis; Synkinesis; Hyperkinesis; Facial Paralysis
Keywords: acquired blepharoptosis; hyperkinesis; synkinesis; facial paralysis; aberrant regeneration syndrome; post-paralysis synkinesis; nonflaccid facial paralysis
MeSH Terms: conditions — Blepharoptosis; Synkinesis; Hyperkinesis; Facial Paralysis | interventions — Oxymetazoline

STUDY DESIGN:
Intervention Model Description: Blinded, randomized, cross-over trial that will analyze and compare the efficacy of oxymetazoline drops alone, oxymetazoline drops adjunct with botulinum toxin, botulinum toxin alone, and no treatment.
Who Masked: Investigator
Masking Description: Participants in the study will be randomized 2:1 to treatment with oxymetazoline 0.1% or the vehicle solution. Randomization schemes were created by a biostatician. This will be stored in a secure database, only accessible to the investigators. Experimental drops and placebo drops will be removed from their labeled boxes and provided to patients with instructions on use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxymetazoline 0.1% ophthalmic drops (Experimental): Patients will use once daily in affected eye. Drops are provided in single use vials.
  Interventions: Drug: Oxymetazoline 0.1% (Pf) Oph Soln Ud
- Preservative free lubricating drops (Placebo Comparator): Patients will use once daily in affected eye. Drops are provided in single use vials.
  Interventions: Other: Preservative free lubricating drops

INTERVENTIONS:
Drug: Oxymetazoline 0.1% (Pf) Oph Soln Ud — Oxymetazoline was initially developed in 1961. It is a direct sympathomimetic, binding directly to alpha-1 and alpha-2 receptors. Currently, it is used as a nasal decongestant, in the treatment of epistaxis, and as a topical treatment for rosacea. Previously, an ophthalmic formulation was used to treat eye redness and irritation as it is FDA approved for the treatment of acquired blepharoptosis. However, this product line was discontinued when in July of 2020, oxymetazoline received Food and Drug Administration approval for treatment of cosmetic blepharoptosis.
  In the treatment of blepharoptosis, oxymetazoline acts on the superior tarsal muscle, Müller's muscle, to elevate the eyelid. The superior tarsal muscle is a sympathetically innervated muscle that is partially responsible for elevating the eyelid. Previous cosmetic studies have shown oxymetazoline can serve as an adjunct to botulinum toxin in patients with acquired blepharoptosis.
  Other Names: Upneeq
  Arms: Oxymetazoline 0.1% ophthalmic drops
Other: Preservative free lubricating drops — Over the counter ophthalmic lubricating drop.
  Other Names: soothe
  Arms: Preservative free lubricating drops

SUMMARY:
After an episode of facial paralysis, as nerves recover, they aberrantly regenerate and send additional branches to the incorrect muscles in addition to the intended muscle. This leads to what is known as Aberrant Regeneration Syndrome, Post-paralysis Synkinesis, or Nonflaccid Facial Paralysis. It is characterized by poor facial symmetry and function, hypertonic facial muscles at rest, and abnormal facial movements. One sequela is acquired blepharoptosis causing a smaller ocular aperture, visual field obstruction, cosmetic deformity, and abnormal periocular spasms. This study aims to evaluate an FDA approved medication for acquired blepharoptosis due to synkinesis/hyperkinesis as an adjunct to treatment.

DETAILED DESCRIPTION:
Broadly, synkinesis is a neuromuscular condition in which voluntary muscle contraction causes simultaneous involuntary contraction of other muscle groups e.g. pursing of the lips causes involuntary closure of the eye. It is a common sequelae of facial nerve paralysis with 55% or more of patients reporting synkinetic facial movement. 2 Additionally, patients may develop hyperkinesis due to continual firing of nerves that have aberrantly regenerated, thereby causing decreased movement due to antagonistic muscle hyperactivity, tightness, spasms, and pain. These together significant affect facial symmetry, aesthetics, and facial function.

While the definitive pathophysiology of synkinesis is still unknown, the most supported theory describes neuronal miswiring (aberrant regeneration theory). It suggests that following injury to the facial nerve and Wallerian degeneration, axons from the facial nucleus in the brainstem regrow and form inappropriate connections to peripheral muscle groups (e.g. a nerve meant to control the orbicularis oris of the mouth connects to the orbicularis oculi of the eye as well). This results in involuntary facial movements during normal expression and can affect all muscles of facial expression.

Furthermore, because of continual facial muscular tone or hypertonicity, this is not only a dynamic process, but a static one as well. Synkinesis and hypertonicity can cause facial asymmetry and a fixed immobile face ("frozen facies) due to opposing muscles constantly contracting and limiting movement. The result can be unaesthetic: the eyes may look smaller, the commissure (corner) of the mouth may look deviated up and out, the nasolabial fold may look deeper, the base of the nose may be deviated, the chin may be twisted or dimpled, and a band may be seen in the neck. This also presents functional limitations, such as difficulties in articulation, biting of the lip/cheek, nasal obstruction, incomplete oral competency with drooling, watering of the eye (epiphora) and in controlling facial expressions. Patients notice pain, tightness, poor facial movement, and difficulty expressing emotions, loss of their smile, and embarrassment. These limitations decrease confidence and ultimately the patient's quality of life.

Our study intends to look specifically at periocular synkinesis with orbicularis oculi muscle hypertonicity resulting in acquired blepharoptosis over time (i.e. drooping of the eyelid). Periocular synkinesis is partial closure of the eye due to inappropriate contraction of the orbicularis oculi muscle during other facial movement. Hypertonicity of the orbicularis oculi muscle results in the static narrowing of the palpebral fissure (acquired blepharoptosis) and may cause visual obstruction, asymmetry, and an aged appearance in the affected eye and can occur with both dynamic movement and static tone (hyperkinesis).

This facial movement disorder has no cure. Treatments are intended to improve facial symmetry, decreased tightness/pain, improve function and improve quality of life. These include facial therapy, chemodenervation injections with neurotoxins, and a variety of surgeries. Patients require multimodal therapy. None of these treatments adequately address the acquired blepharoptosis from chronic hyperkinesis and synkinesis.

Oxymetazoline was initially developed in 1961. It is a direct sympathomimetic, binding directly to alpha-1 and alpha-2 receptors. Currently, it is used as a nasal decongestant, in the treatment of epistaxis, and as a topical treatment for rosacea. Previously, an ophthalmic formulation was used to treat eye redness and irritation as it is FDA approved for the treatment of acquired blepharoptosis. However, this product line was discontinued when in July of 2020, oxymetazoline received Food and Drug Administration approval for treatment of cosmetic blepharoptosis.

In the treatment of blepharoptosis, oxymetazoline acts on the superior tarsal muscle, Müller's muscle, to elevate the eyelid. The superior tarsal muscle is a sympathetically innervated muscle that is partially responsible for elevating the eyelid. 5 Previous cosmetic studies have shown oxymetazoline can serve as an adjunct to botulinum toxin in patients with acquired blepharoptosis. However, no study has been performed evaluating oxymetazoline's efficacy as an adjunct to botulinum toxin in patients with acquired blepharoptosis secondary to hypertonicity and synkinesis.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Primary diagnosis of nonflaccid facial paralysis (aberrant regeneration syndrome) and acquired blepharoptosis.

Exclusion Criteria:

1. Patients under the age of 18
2. Patients on cardiac glycosides
3. Patients on MAO inhibitors
4. Patients with angle closure glaucoma
5. Patients who experience asymmetrical eye opening due to weakness (e.g. lagophthalmos).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-01-08 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference from baseline to end of study in Sunnybrook Grading Score | 6 months
  Clinician-graded outcome measure
Difference from baseline to end of study Synkinesis Assessment Questionnaire | 6 months
  Patient reported outcome measure
Difference from baseline to end of study in Facial Disability Index | 6 months
  Disease-specific quality of life measure

SECONDARY OUTCOMES:
Difference in MRD-1 from baseline to when medication is being used | 6 months
  Objective assessment of eyelid position relative to the pupillary light reflex as measured by clinician
Difference in palpebral height from baseline to when medication is being used | 6 months
  Width of ocular aperture from upper to lower eyelid

CONTACTS AND LOCATIONS:
Overall Officials: Jessyka Lighthall, MD, Principal Investigator — Penn State Health
Locations (1):
- M.S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No